CLINICAL TRIAL: NCT05703867
Title: Interventional Study of Transpalpebral Microcurrent Stimulation for the Improvement of Visual Acuity in Patients With Macular Degeneration
Brief Title: Transpalpebral Microcurrent Stimulation for the Improvement of Visual Acuity in Patients With Macular Degeneration
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Jarding, John, OD (Individual)
Collaborators: Professor Timothy Jackson, King's College (Unknown); i-Lumen Scientific, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OL101
Record Dates: First submitted 2023-01-20; First posted 2023-01-30 (Actual); Last update posted 2023-01-31 (Actual); Status verified 2023-01

CONDITIONS: Age-Related Macular Degeneration; Nonexudative Age-related Macular Degeneration
MeSH Terms: conditions — Macular Degeneration

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- Active microcurrent therapy (Experimental)
  Interventions: Device: Active microcurrent therapy

INTERVENTIONS:
Device: Active microcurrent therapy — Non-invasive transpalpebral microcurrent therapy delivery to the upper and lower eyelids

SUMMARY:
The goal of this clinical trial is to evaluate the effectiveness of transpalpebral microcurrent stimulation as a therapy for dry age-related macular degeneration.

Participants are assessed at baseline for visual acuity and treated for 4 consecutive days for a total of 8 sessions (2 per day) with microcurrent stimulation. A follow-up visit is conducted to evaluate the participant and collect follow-up visual acuity.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged at least 50 years with dry AMD in at least one eye

Exclusion Criteria:

* Eye diseases other than dry AMD
* Implanted electrical devices
* Seizure disorders

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 404 (Actual)
Dates: Start 1998-01 (Actual); Primary Completion 1999-12 (Actual); Study Completion 1999-12 (Actual)

PRIMARY OUTCOMES:
Mean logMAR BCVA | Week 1
  Mean logarithm of the minimum angle of resolution (logMAR) best-corrected visual acuity (BCVA) following the last treatment

SECONDARY OUTCOMES:
Proportion of improved, stable or worsened BCVA | Week 1
  Proportion of eyes with improved, stable or worsened BCVA, and BCVA with both eyes open